CLINICAL TRIAL: NCT05132192
Title: Outcomes of Surgical Strategies for Living Donor Liver Transplantation to Patients With Portal Vein Thrombosis
Brief Title: Living Donor Liver Transplantation to Patients With Portal Vein Thrombosis
Status: Completed | Type: Observational
Sponsor: Elvan Onur Kirimker (Other)
Collaborators: Ankara University (Other); Ankara Guven Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Elvan Onur Kirimker, Attending surgeon at Dept of Surgery, Ankara University
Organization: Ankara University (Other)
Other Study IDs: PVT-LDLT-ANK
Record Dates: First submitted 2021-10-28; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Portal Vein Thrombosis; Liver Transplant; Complications
Keywords: Liver transplantation; Portal vein thrombosis; Thrombectomy; Doppler flowmeter
MeSH Terms: interventions — Thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PVT: Patients with pretransplant portal vein thrombosis
  Interventions: Procedure: living donor liver transplantation; Procedure: Thrombectomy or interposition graft
- non-PVT: Patients without pretransplant portal vein thrombosis
  Interventions: Procedure: living donor liver transplantation

INTERVENTIONS:
Procedure: living donor liver transplantation — Living donor liver transplantation
Procedure: Thrombectomy or interposition graft — Portal flow restoration due to PVT in any manner
  Groups: PVT

SUMMARY:
Data of demographic, clinical, laboratory and imaging studies of living donor liver transplantation (LDLT) recipients from two transplant centers were collected. Survival and morbidity rates between patients with and without portal vein thrombosis (PVT) were compared. Risk factors of mortality in the setting of PVT were identified. Intraoperative portal flow measurements were compared before and after portal flow restoration.

DETAILED DESCRIPTION:
LDLTs performed in two experienced centers (Ankara University Ibn-i Sina Hospital and Ankara Güven Hospital) between January 2013 and February 2020 were evaluated and included in the cohort study. Deceased donor liver transplants and pediatric transplants (deceased or living) were excluded from the study.

Data relating to this study including patient history, preoperative laboratory and imaging test results, reports of surgical procedures or interventions, intraoperative anesthesia records, post-operative laboratory trends, and postoperative complications were extracted from the computer-based data management system and prospectively maintained in transplant databases in both centers. Recipients of LDLT were divided in two groups according to the presence or absence of PVT.

Portal flow measurements were recorded with VeriQ (Medistim ASA, Oslo, Norway) Doppler flowmeter device in one of the centers later in the study period.

The follow-up and recordings of the patients were maintained in the outpatient clinics of the two centers.

The most serious complication experienced by each patient was recorded according to the Clavien-Dindo classification Primary outcome of the current study was the survival rates of patients with and without PVT Secondary outcomes of the study included morbidity in patients with and without PVT after LDLT, risk factors of mortality after LDLT to patients with PVT and comparison of intraoperative portal flow measurements between patients with and without PVT

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent liver transplantation

Exclusion Criteria:

* Pediatric liver transplants
* Deceased donor liver transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients that who underwent living donor liver transplantation in the study period in the two centers
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Survival | Time (days) from post transplant day1 to post transplant1 year
  Posttransplant survival time

SECONDARY OUTCOMES:
Complications | From posttransplant day1 to post-transplant 30th day
  Highest grade of complication after LDLT according to Dindo-Clavien Classification
Flow | Intraoperatively twice: before recipient hepatectomy (portal flow of diseased liver ) and at the end of transplantation procedure
  Intraoperative portal flow measurements (ml/min) of diseased liver and transplanted liver with Doppler flowmeter

CONTACTS AND LOCATIONS:
Overall Officials: Elvan O Kirimker, MD, Principal Investigator — Ankara University

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

REFERENCES:
- [Background] Conzen KD, Pomfret EA. Liver transplant in patients with portal vein thrombosis: Medical and surgical requirements. Liver Transpl. 2017 Oct;23(S1):S59-S63. doi: 10.1002/lt.24856. No abstract available. PMID 28834305
- [Background] Yerdel MA, Gunson B, Mirza D, Karayalcin K, Olliff S, Buckels J, Mayer D, McMaster P, Pirenne J. Portal vein thrombosis in adults undergoing liver transplantation: risk factors, screening, management, and outcome. Transplantation. 2000 May 15;69(9):1873-81. doi: 10.1097/00007890-200005150-00023. PMID 10830225
- [Background] Ravaioli M, Zanello M, Grazi GL, Ercolani G, Cescon M, Del Gaudio M, Cucchetti A, Pinna AD. Portal vein thrombosis and liver transplantation: evolution during 10 years of experience at the University of Bologna. Ann Surg. 2011 Feb;253(2):378-84. doi: 10.1097/SLA.0b013e318206818b. PMID 21183851
- [Background] Zanetto A, Rodriguez-Kastro KI, Germani G, Ferrarese A, Cillo U, Burra P, Senzolo M. Mortality in liver transplant recipients with portal vein thrombosis - an updated meta-analysis. Transpl Int. 2018 Dec;31(12):1318-1329. doi: 10.1111/tri.13353. Epub 2018 Oct 23. PMID 30230053
- [Background] Qi X, Dai J, Jia J, Ren W, Yang M, Li H, Fan D, Guo X. Association between portal vein thrombosis and survival of liver transplant recipients: a systematic review and meta-analysis of observational studies. J Gastrointestin Liver Dis. 2015 Mar;24(1):51-9, 4 p following 59. doi: 10.15403/jgld.2014.1121.qix. PMID 25822434
- [Background] Hibi T, Nishida S, Levi DM, Selvaggi G, Tekin A, Fan J, Ruiz P, Tzakis AG. When and why portal vein thrombosis matters in liver transplantation: a critical audit of 174 cases. Ann Surg. 2014 Apr;259(4):760-6. doi: 10.1097/SLA.0000000000000252. PMID 24299686